CLINICAL TRIAL: NCT05955183
Title: Phase-1, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD5055 Following Single and Multiple Oral Doses in Japanese and Chinese Healthy Volunteers.
Brief Title: Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD5055 in Japanese and Chinese Healthy Volunteers..
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: D8960C00005
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Healthy Participants
Keywords: Single ascending dose (SAD)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD5055 (Active Comparator): Participants will orally receive AZD5055.
  Interventions: Drug: AZD5055; Drug: Placebo
- Placebo (Placebo Comparator): Participants will orally receive placebo.
  Interventions: Drug: AZD5055; Drug: Placebo

INTERVENTIONS:
Drug: AZD5055 — AZD5055 will be given orally to randomized participants as per the arm they are assigned.
Drug: Placebo — Placebo will be given orally to randomized participants as per the arm they are assigned.

SUMMARY:
This study will evaluate the pharmacokinetics (PK), pharmacodynamics (PD), safety, and tolerability of AZD5055 after single and multiple doses, orally administered in healthy Japanese and Chinese participants.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts:

1. Part 1 in single ascending dose (SAD)
2. Multiple dose Eligible Japanese and Chinese participants will be randomized to receive oral dose of either AZD5055 or placebo.

The study will comprise of:

* A Screening Period of maximum 28 days.
* A Treatment Period during which participants will be resident at the Clinical Unit from the day before investigational medicinal product (IMP) administration until at least 72 hours after IMP administration.
* A Follow-up Visit within 7 ± 1 (for Part 1) and 15 ± 1 (for Part 2) days after the last IMP dose.

For the SAD part of the study, each participant will be involved in the study for 5 to 6 weeks.

For the multiple dose part of the study, each participant will be involved in the study for 7 to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* For Chinese subjects only:

  1. Participant was born in greater China, including Hong Kong, Macau, and Taiwan.
  2. Participant has 2 Chinese biological parents and 4 Chinese grandparents as confirmed by interview.
  3. Participant did not live outside of greater China for more than 10 years at the time of the Screening Period.
* For Japanese subjects only:

  1. Participant was born in Japan.
  2. Participant has 2 Japanese biological parents and 4 Japanese grandparents as confirmed by the interview.
  3. Participant did not live outside of Japan for more than 10 years at the time of the Screening Period.
* Females must have a negative pregnancy test at the Screening Visit, must not be lactating and must be of non-childbearing potential.
* Males must adhere to the contraception methods.
* Have a Body mass index between 18 and 30 kg/m2 inclusive.

Exclusion Criteria:

* History of any clinically significant disease or disorder which may either put the participant at risk because of participation in the study or influence the results or the participant's ability to participate in the study.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of study drug.
* Any abnormal laboratory values.
* Participants with chronic infections (eg, urinary tract infection) or who are at increased risk of infection.
* History of cancer within the last 10 years.
* History of osteoporosis, osteomalacia, Paget's disease of the bone, thyrotoxicosis, rheumatoid arthritis, Cushing's disease, or a pathological fracture.
* History of traumatic fracture within 6 months of the Screening Visit.
* Participants will be excluded if

  1. In premenopausal women, men less than 50 years of age: Z-scores ≤ -2.0.
  2. In postmenopausal women and men aged 50 years and older: T-score ≤ -2.5.
* Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results.
* Abnormal vital signs.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting electrocardiogram (ECG) and any clinically important abnormalities in the 12 lead ECG.
* History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5055.
* Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 30 days (or 5 half-lives, whichever is the longest) of the first administration of study drug in this study.
* Has a body temperature of > 37.7°C.
* Untreated Tuberculosis or a positive result for the Interferon gamma release assay.
* Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody, and Human immunodeficiency virus.
* History of Gilbert's syndrome.
* History of muscle disease or rhabdomyolysis.
* Plasma donation within one-month of the Screening Visit or any blood donation/blood loss more than 500 mL.
* Positive screen for drugs of abuse (excluding cannabis) at Screening.
* Current smokers who smoke > 20 cigarettes/e-cigarettes/pipes per week.
* Use of drugs with enzyme inducing properties.
* Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, mega dose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks or 5 half-lives of the medication, whichever is longer, prior to the first administration of study drug.
* Excessive intake of caffeine-containing drinks or food.
* Study participation by an AstraZeneca or Clinical Unit employee directly involved in the study.
* Participants who have previously received AZD5055.
* Participants who have minor medical complaints which can interfere with the study data.
* Participants who are vegans or have medical dietary restrictions.
* Participants who cannot communicate reliably with the Investigator.
* Vulnerable participants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Until Follow-up (Day 7 ± 1 for Part 1 and Day 15 ± 1 for Part 2).
  The safety and the tolerability after single and multiple doses of AZD5055 in healthy Japanese and Chinese participants will be evaluated.

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) | Day 1 to Day 3 (Part 1) and Day 1 to Day 10 (Part 2)
  The Cmax after administration of single and multiple doses of AZD5055 in healthy Japanese and Chinese participants will be evaluated.
Area under plasma concentration-time curve from time 0 to infinity (AUCinf) | Day 1 to Day 3 (Part 1) and Day 1 to Day 10 (Part 2)
  The AUCinf after administration of single and multiple doses of AZD5055 in healthy Japanese and Chinese participants will be evaluated.
Area under plasma concentration-curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 to Day 3 (Part 1) and Day 1 to Day 10 (Part 2)
  AUClast after administration of single and multiple doses of AZD5055 in healthy Japanese and Chinese participants will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States